CLINICAL TRIAL: NCT03772574
Title: Preoxygenation Using THRIVE and Facemask Oxygenation in Parturients
Brief Title: Preoxygenation Using THRIVE Versus Facemask in Parturients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H18-02855
Record Dates: First submitted 2018-12-08; First posted 2018-12-11 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Preoxygenation
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE (Experimental): THRIVE preoxygenation (tidal volume breathing with the OptiFlow system applied at 100% oxygen).
  Interventions: Device: THRIVE preoxygenation
- Facemask (Active Comparator): Facemask preoxygenation (tidal volume breathing via a face mask set at 100% oxygen).
  Interventions: Device: Facemask preoxygenation

INTERVENTIONS:
Device: Facemask preoxygenation — Standard facemask preoxygenation
  Arms: Facemask
Device: THRIVE preoxygenation — Preoxygenation using transnasal humidified rapid insufflation ventilatory exchange (THRIVE).
  Other Names: THRIVE
  Arms: THRIVE

SUMMARY:
This study aims to determine the duration for pre-oxygenation using THRIVE and facemask for parturients.

DETAILED DESCRIPTION:
We aim to determine the duration required for THRIVE and facemask preoxygenation in parturients for them to achieve ETO2 >90%.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients ≥36 weeks gestation.
* Non-laboring patients admitted for elective Cesarean delivery under neuraxial anesthesia or induction of labor.
* American Society of Anesthesiologists (ASA) class 2.

Exclusion Criteria:

* Any medical conditions that are likely to affect gas exchange.
* Obstructed nasal passage.
* Unable to tolerate a tight fitting facemask.
* Body Mass Index ≥40 kg/m2.
* Patients who are in active labor (i.e. cervical dilation ≥4cm).
* Patients who are unable to give informed consent.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 91 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD MMSc, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Au K, Shippam W, Taylor J, Albert A, Chau A. Determining the effective pre-oxygenation interval in obstetric patients using high-flow nasal oxygen and standard flow rate facemask: a biased-coin up-down sequential allocation trial. Anaesthesia. 2020 May;75(5):609-616. doi: 10.1111/anae.14995. Epub 2020 Feb 11. PMID 32048278

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 91 patients provided informed consent in order to reach the recruitment goal of 80 patients. This is the reason for the discrepancy mentioned in the comments.
Groups:
- Standard Facemask: Facemask preoxygenation (tidal volume breathing via a face mask set at 100% oxygen).
  Facemask preoxygenation: Standard facemask preoxygenation
- THRIVE and Facemask: THRIVE preoxygenation (tidal volume breathing with the OptiFlow system applied at 100% oxygen). Facemask used to minimize air entrainment
  THRIVE preoxygenation: Preoxygenation using transnasal humidified rapid insufflation ventilatory exchange (THRIVE).
Period: Overall Study
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
Started | 42 | 25 | 24
Completed | 40 | 20 | 20
Not Completed | 2 | 5 | 4
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Discomfort | 0 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask | Total
Number analyzed (Participants) | 40 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (4.3) | 35 (4.1) | 35 (4.4) | 35.3 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 20 | 20 | 80
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 40 | 20 | 20 | 80
Gravidity [Median (Inter-Quartile Range); unit: Pregnancies] | 2 [2 to 3] | 2 [2 to 4] | 2 [2 to 2] | 2 [2 to 3]
Parity [Median (Inter-Quartile Range); unit: births] | 1 [0 to 1] | 1 [0 to 1] | 1 [0 to 1] | 1 [0 to 1]
Gestational age [Mean (Standard Deviation); unit: weeks] | 38.6 (1.0) | 38.7 (1.1) | 39.1 (0.6) | 38.8 (0.92)
Baseline respiratory rate [Mean (Standard Deviation); unit: breaths/min] | 11.9 (3.7) | 14.5 (4.1) | 13.3 (3.1) | 12.9 (3.8)
Baseline End Tidal Oxygen (ETO2) [Mean (Standard Deviation); unit: Percent of oxygen in expired breath] | 15.7 (1.2) | 15.7 (0.9) | 15.8 (1.0) | 15.7 (1.1)
Baseline Heart Rate [Mean (Standard Deviation); unit: bpm] | 74.4 (10.8) | 76.1 (9.7) | 75.2 (13.9) | 75.1 (11.3)
Baseline Oxygen Saturation (SPO2) [Mean (Standard Deviation); unit: percent of hemoglobin carrying oxygen] | 98.0 (1.5) | 98.4 (1.4) | 98.5 (1.4) | 98.2 (1.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (3.7) | 29.5 (4.8) | 30.4 (3.8) | 29.5 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Preoxygenation Duration
Description: Duration to achieve EtO2 >=90% after tidal volume breathing using THRIVE and facemask pre-oxygenation.
Time Frame: Maximum 8 minutes
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
Number analyzed (Participants) | 40 | 20 | 20
minutes | 3.6 [3.3 to 6.7] | NA [NA to NA] — A value could not be entered, as the longest possible preoxygenation time allotment (8 minutes) was insufficient to produce an EI90 | NA [NA to NA] — A value could not be entered, as the longest possible preoxygenation time allotment (8 minutes) was insufficient to produce an EI90

2. Secondary Outcome: Proportion to Reach End Tidal Oxygen (ETO2) of 90 Percent at 3 Minutes
Time Frame: 3 minutes of pre-oxygenation
Population: Patients selected to receive 3 minutes of pre-oxygenation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
Number analyzed (Participants) | 14 | 2 | 1
Participants | 10 | 0 | 0

3. Secondary Outcome: Proportion to Reach EtO2 of 90 Percent at 4 Minutes
Time Frame: 4 minutes of preoxygenation
Population: Patients assigned to recieve 4 minutes of pre-oxygenation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
Number analyzed (Participants) | 26 | 3 | 5
Participants | 26 | 2 | 4

4. Secondary Outcome: Proportion to Reach EtO2 of 90 Percent at 5 Minutes
Time Frame: 5 minutes of preoxygenation
Population: Patients assigned to receive 5 minutes of pre-oxygenation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
Number analyzed (Participants) | 0 | 1 | 1
Participants | 0 | 0 | 0

5. Secondary Outcome: Proportion to Reach EtO2 of 90 Percent at 6 Minutes
Time Frame: 6 minutes of preoxygenation
Population: Patients assigned to receive 6 minutes of preoxygenation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
Number analyzed (Participants) | 0 | 1 | 1
Participants |  | 0 | 0

6. Secondary Outcome: Proportion to Reach EtO2 of 90 Percent at 7 Minutes
Time Frame: 7 minutes of preoxygenation
Population: Patients assigned to receive 7 minutes of preoxygenation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
Number analyzed (Participants) | 0 | 1 | 1
Participants | 0 | 0 | 0

7. Secondary Outcome: Proportion to Reach EtO2 of 90 Percent at 8 Minutes
Time Frame: 8 minutes of preoxygenation
Population: patients assigned to receive 8 minuets of pre-oxygenation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
Number analyzed (Participants) | 0 | 12 | 11
Participants | 0 | 1 | 5

8. Secondary Outcome: Comfort Score
Description: Patients were asked to rate their comfort with the device on a 5 point Likert Scale: (1=completely uncomfortable, 2=slightly uncomfortable, 3=neutral, 4=slightly comfortable, 5= completely comfortable)
Time Frame: 1 minute after data collection
Measure: Median (Inter-Quartile Range); unit: Likert Score
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
Number analyzed (Participants) | 40 | 20 | 20
Likert Score | 4 [2 to 5] | 4 [2 to 4] | 4 [3 to 5]

9. Secondary Outcome: Acceptability Score
Description: Acceptability was measured with a 5-point Likert Score (1= unacceptable, 2=slightly unacceptable,3=neutral, 4=slightly acceptable, 5=acceptable).
Time Frame: 1 minute after data collection
Measure: Median (Inter-Quartile Range); unit: Likert Score
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
Number analyzed (Participants) | 40 | 20 | 20
Likert Score | 5 [4 to 5] | 4.5 [3.75 to 5] | 5 [5 to 5]

ADVERSE EVENTS:
Time Frame: 7 months
Description: Patients are not at risk of any adverse events other than some discomfort during preoxygentaion. The study team was careful to avoid complications of pressure related damage to the lungs, by limiting the period of time patients were exposed to high flow oxygen to 8 minutes.
Arm/Group | Standard Facemask | THRIVE | THRIVE and Facemask
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/42 | 0/25 | 0/24

LIMITATIONS AND CAVEATS:
Our results are specific to healthy parturients using standard facemasks, or a high oxygen flow rate of 50L/min, and cannot be generalized to other techniques or populations. 9 parturients left the study due to discomfort, which may bias outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT03772574/Prot_SAP_000.pdf